CLINICAL TRIAL: NCT04938700
Title: Study on the Correlation Between Intestinal Microecology and Allergic Diseases in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Provincial Hospital of TCM (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Zibo Central Hospital (Other Government); The First People's Hospital of Huzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-276
Record Dates: First submitted 2021-06-03; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-05

CONDITIONS: Rhinitis, Allergic; Asthma; Dermatitis, Atopic; Urticaria
Keywords: Probiotics; Hypersensitivity; Gastrointestinal Microbiome; immunity
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Dermatitis, Atopic; Urticaria; Hypersensitivity | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics intervention group (Experimental): children with definitive diagnosis of allergic rhinitis, asthma，atopic dermatitis and chronic urticaria were enrolled, each with 25 cases. 2) collect manure application of 16s rDNA probe hybridization technique to analyze the fecal flora, and compared with clinical symptoms rating scale and serum sIgE, IgG4 correlation analysis (3) application of probiotic intervention and conventional drugs, again in 3 months, 6 months after collecting dung is used to detect the intestinal flora in children with its correlation with clinical symptoms change were observed.
  Interventions: Drug: probiotics; Drug: conventional medical treatment
- Contrast group (Active Comparator): children with definitive diagnosis of allergic rhinitis, asthma，atopic dermatitis and chronic urticaria were enrolled, each with 25 cases. 2) collect manure application of 16s rDNA probe hybridization technique to analyze the fecal flora, and compared with clinical symptoms rating scale and serum sIgE, IgG4 correlation analysis (3) application of conventional drugs, again in 3 months, 6 months after collecting dung is used to detect the intestinal flora in children with its correlation with clinical symptoms change were observed.
  Interventions: Drug: conventional medical treatment

INTERVENTIONS:
Drug: probiotics — Probiotics as granules can be used for infants and adolescents
  Other Names: conventional medical treatment
  Arms: Probiotics intervention group
Drug: conventional medical treatment — Treatment for allergic diseases includes anti-allergic drugs, nasal spray hormones, inhaled hormones, external hormones, etc

SUMMARY:
Allergic diseases, including allergic reactions of respiratory tract and skin, are often triggered by mast cell degranulation mediated by allergen-specific IgE and chronic inflammation of target organs, which are involved in a variety of immune cells and inflammatory factors. Recent studies have shown that intestinal immunity is closely related to immune responses to various diseases. Intestinal microecology influences the occurrence and regression of various diseases by regulating the growth, differentiation and maturation of various immune cells. Probiotics are widely used in children with allergies. This study aims to analyze the correlation between the intestinal microecology of children with rhinitis/asthma, eczema and urticaria and the clinical manifestations of the patients. By observing the influence of probiotics intervention on clinical symptoms and changes in intestinal microecology, the influence of intestinal microecology on children's allergic diseases was clarified. Study protocol: 1) children with definitive diagnosis of allergic rhinitis, asthma，atopic dermatitis and chronic urticaria were enrolled, each with 50 cases. 2) collect manure application of 16s rDNA probe hybridization technique to analyze the fecal flora, and compared with clinical symptoms rating scale and serum sIgE, IgG4 correlation analysis (3) application of probiotic intervention or conventional drug intervention, again in 3 months, 6 months after collecting dung is used to detect the intestinal flora in children with its correlation with clinical symptoms change were observed.

DETAILED DESCRIPTION:
1. Fifty children（0-14years）with clear diagnosis of allergic rhinitis, asthma，atopic dermatitis and chronic urticaria were selected.
2. Feces were collected for analysis of fecal flora by 16S rDNA probe hybridization, and the correlation between the fecal flora and clinical symptom scoring scale, serum sIgE and IgG4 was analyzed.
3. Using probiotics intervention or conventional symptomatic drug intervention, the feces of the children were collected again after 3 months and 6 months for intestinal flora detection, and the correlation with clinical symptoms was observed. Probiotics for granules a blunt and can be used for infants and young children and adolescents, conventional drugs within 2 years old infant antihistamines for children drops, nasal drops and atomization inhalation antiasthmatic, 2-5 years of age can contain montelukast sodium chewing tablets, children over the age of five, including inhaled corticosteroids, oral antihistamines and montelukast sodium chewing tablets and expectorant drugs.
4. Inclusion criteria: patients with allergic rhinitis, asthma, atopic dermatitis or urticaria aged 0-14 years with elevated serum total IgE were clinically diagnosed as allergic patients.
5. Exclusion criteria: patients who withdrew due to treatment intolerance or other reasons during the treatment process.

The study involved children, but the feces were collected and measured in vitro, which was harmless to children.

ELIGIBILITY:
Inclusion Criteria:

* Elevated serum total IgE in patients with allergic rhinitis, asthma, atopic dermatitis, and chronic urticaria aged 0-14 years

Exclusion Criteria:

* Patients who withdraw during treatment due to treatment intolerance or other reasons

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The distribution and quantity of intestinal flora（Determination of fecal microecology by 16S rDNA probe hybridization） | 1 year
  The changes of intestinal flora before and after the application of probiotics;Difference of intestinal flora distribution between control group and intervention group.Determination of fecal microecology by 16S rDNA probe hybridization. It included intestinal flora balance, flora diversity, bacterial strain number and pathogenic bacteria detection.
Clinical symptoms rating scale-Allergic rhinitis symptom rating scale （TNSS+TNNSS） | 1 year
  The changes of clinical symptoms rating scale before and after the application of probiotics; Difference of clinical symptoms rating scale between control group and intervention group.Allergic rhinitis symptom rating scale TNSS+TNNSS，the minimum value is 1，the maximum value is 4，and higher scores mean a worse outcome
Clinical symptoms rating scale-Asthma Control Score Scale (ACT) | 1 year
  The changes of clinical symptoms rating scale before and after the application of probiotics; Difference of clinical symptoms rating scale between control group and intervention group.Asthma Control Score Scale (ACT)，the minimum value is 1，the maximum value is 5，and higher scores mean a worse outcome
Clinical symptoms rating scale-Dermatology Quality of Life Indicators Inventory (DLQI) | 1year
  The changes of clinical symptoms rating scale before and after the application of probiotics; Difference of clinical symptoms rating scale between control group and intervention group.Dermatology Quality of Life Indicators Inventory (DLQI)：the minimum value is 0，the maximum value is 3，and higher scores mean a worse outcome.
sIgE | 1 year
  The changes of sIgE（IU/ml） before and after the application of probiotics; Difference of sIgE between control group and intervention group
IgG4 | 1 year
  The changes of IgG4（U/ml） before and after the application of probiotics; Difference of IgG4 between control group and intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Wang, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital，School of Medicine，Zhejiang University, Hangzhou, Zhejiang, China